CLINICAL TRIAL: NCT04418661
Title: A Phase 1/2, Open-label, Multicenter, Dose Escalation and Dose Expansion Study of SAR442720 in Combination With Other Agents in Participants With Advanced Malignancies
Brief Title: Safety and Efficacy Study of Vociprotafib (SAR442720) in Combination With Other Agents in Advanced Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision not related to any safety concern
Sponsor: Sanofi (Industry)
Collaborators: Revolution Medicines, Inc. (Industry); Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TCD16210; U1111-1244-2555 (Registry Identifier: ICTRP); TCD16210 (Other: Sanofi Identifier); 2020-000436-22 (EudraCT Number)
Record Dates: First submitted 2020-05-29; First posted 2020-06-05 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — pembrolizumab; adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1- SAR442720 140 mg BIW + Pembrolizumab (Experimental): Participants were administered SAR442720 140 milligram (mg) orally twice a week (BIW) on Days 1 and 4 along with pembrolizumab 200 mg via intravenous (IV) infusion once every 3 weeks (Q3W) in 21-day cycles until disease progression, unacceptable adverse events (AEs), or the participant's or investigator's decision to stop the treatment.
  Interventions: Drug: Vociprotafib; Drug: Pembrolizumab
- Part 1- SAR442720 200mg BIW + Pembrolizumab (Experimental): Participants were administered SAR442720 200 mg orally BIW on Days 1 and 2 along with pembrolizumab 200 mg via IV infusion Q3W in 21-day cycles until disease progression, unacceptable AEs, or the participant's or investigator's decision to stop the treatment.
  Interventions: Drug: Vociprotafib; Drug: Pembrolizumab
- Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%) (Experimental): Participants with programmed death-ligand 1 (PD-L1) tumor proportion score (TPS)>=50% non-small cell lung cancer (NSCLC) were administered SAR442720 200 mg orally BIW on Days 1 and 2 in 21-day cycles along with an IV infusion of pembrolizumab 200 mg on Q3W (21 days cycle) or 400 mg once in every 6 weeks (Q6W) (42 days cycle) until disease progression, unacceptable AEs, consent withdrawal, or the participant's or investigator's decision to stop the treatment.
  Interventions: Drug: Vociprotafib; Drug: Pembrolizumab
- Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%) (Experimental): Participants with PDL1 TPS 1% - 49% NSCLC were administered SAR442720 200 mg orally BIW on Days 1 and 2 in 21-day cycles along with an IV infusion of pembrolizumab 200 mg on Q3W (21 days cycle) or 400 mg Q6W (42 days cycle) until disease progression, unacceptable AEs, consent withdrawal, or the participant's or investigator's decision to stop the treatment.
  Interventions: Drug: Vociprotafib; Drug: Pembrolizumab
- Part 3A- SAR442720 100mg BIW + Adagrasib (Experimental): Participants were administered SAR442720 100 mg orally BIW on Days 1 and 2 along with adagrasib 400 mg orally twice daily (BID) in 21-day cycles until disease progression, unacceptable AEs, consent withdrawal, or the participant's or investigator's decision to stop the treatment.
  Interventions: Drug: Vociprotafib; Drug: Adagrasib
- Part 4- SAR442720 200mg + Pembrolizumab (Experimental): Participants were administered SAR442720 200 mg orally BIW on Days 1 and 2 in 21-day cycles (as tablet during the first cycle and as capsule from Cycle 2) along with an IV infusion of pembrolizumab 200 mg Q3W (21-day cycle)or 400 mg Q6W (42-day cycle) until disease progression, unacceptable AEs, consent withdrawal, or the participant's or investigator's decision to stop the treatment.
  Interventions: Drug: Vociprotafib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Vociprotafib — Pharmaceutical form: Varies Route of administration: Varies
  Other Names: SAR442720, RMC-4630
Drug: Pembrolizumab — Pharmaceutical form:Sterile Lyophilized powder for reconstitution Route of administration: Infusion
  Arms: Part 1- SAR442720 140 mg BIW + Pembrolizumab; Part 1- SAR442720 200mg BIW + Pembrolizumab; Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%); Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%); Part 4- SAR442720 200mg + Pembrolizumab
Drug: Adagrasib — Pharmaceutical form:Sterile Tablet Route of administration: Oral
  Arms: Part 3A- SAR442720 100mg BIW + Adagrasib

SUMMARY:
Primary Objectives:

* Part 1
* To characterize the safety and tolerability of SAR442720 in combination with pembrolizumab in participants with advanced solid tumors.
* To define the MTD and RP2D for the combination of SAR442720 and pembrolizumab in participants with solid tumors.
* Part 2
* To determine the anti-tumor activity of SAR442720 in combination with pembrolizumab.
* Part 3A
* To define the MTD and RP2D for the combination of SAR442720 and adagrasib in participants with KRAS G12C NSCLC
* To characterize the safety and tolerability of SAR442720 in combination with adagrasib in participants with KRAS G12C NSCLC
* Part 3B
* To determine the anti-tumor activity of SAR442720 in combination with adagrasib in participants with KRAS G12C NSCLC
* Part 4
* To evaluate the impact of food on the PK of SAR442720 when dosed with pembrolizumab.
* To evaluate the impact of the formulations (formulation 1 and formulation 2) on the PK of SAR442720 when dosed with pembrolizumab.

Secondary Objectives:

* Part 1
* To assess the PK of SAR442720 with pembrolizumab, and the PK of pembrolizumab with SAR442720.
* To estimate the anti-tumor effects of SAR442720 with pembrolizumab.
* Part 2
* To assess the safety profile of SAR442720 combined with pembrolizumab.
* To assess other indicators of anti-tumor activity.
* To assess the PK of SAR442720 with pembrolizumab, and the PK of pembrolizumab with SAR442720.
* Part 3A
* To characterize the PK of SAR442720 with adagrasib, and the PK of adagrasib with SAR442720.
* To estimate the anti-tumor effects of SAR442720 with adagrasib
* Part 3B
* To assess the safety profile of SAR442720 with adagrasib in participants with KRAS G12C NSCLC.
* To assess other indicators of anti-tumor activity.
* To assess the PK of SAR442720 with adagrasib, and the PK of adagrasib with SAR442720.
* Part 4
* To assess the safety and tolerability of SAR442720 formulations with pembrolizumab
* To estimate the anti-tumor effects of SAR442720 with pembrolizumab.

DETAILED DESCRIPTION:
This open label Phase 1 multicenter study was designed to evaluate the safety and maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of SAR442720 in combination with pembrolizumab in participants with solid tumors in Part 1.

In Part 2, in the expansion cohort (Cohort A) we assessed the antitumor activity and safety of SAR442720 combined with pembrolizumab in participants with metastatic 1L lung cancer.

In Part 3, we evaluated the safety, MTD, RP2D and antitumor activity of SAR442720 in combination with adagrasib in participants with lung cancer and KRAS G12C mutation.

In Part 4, we evaluated the impact of the formulations (formulation 1 and formulation 2) and of the food on the PK of SAR442720 when dosed in combination with pembrolizumab. The expected duration of study intervention for participants may vary, based on progression date; median expected duration of study per participant was estimated to be about 10 months in Part 1, Part 3 and Part 4 (up to 1 month for screening, a median of 6 months for treatment, and a median of 3 months for long term follow-up) and in Part 2 16 months (up to 1 month for screening, a median of 12 months for treatment and a median of 3 months for long term follow up.)

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥ 18 years of age.
* Histologically proven diagnosis of advanced solid tumors.
* Participants must have one or more of the following molecular aberrations (Part 1): KRAS mutations and amplifications, BRAF Class 3 mutations, or NF1 LOF mutations.
* Participants must have following molecular aberration (Part 3A and 3B): - KRAS G12C mutation.
* At least 1 measurable disease per RECIST 1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Woman of childbearing potential must agree to follow contraceptive guidance.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Predicted life expectancy <3 months.
* Primary central nervous system (CNS) tumors.
* Symptomatic or impending cord compression. Stable CNS disease was allowed.
* History of cerebrovascular stroke or transient ischemic attack within previous 6 months.
* Prior solid organ or hematologic transplant.
* History or current retinal pigment epithelial detachment (RPED), central serous retinopathy, retinal vascular occlusion (RVO), neovascular macular degeneration.
* Any clinically significant cardiac disease.
* Active, known or suspected autoimmune disease.
* History of or current interstitial lung disease or pneumonitis.
* Receipt of a live-virus vaccination within 28 days, viral vaccine that do not contain live virus within 7 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.
* Known infection with human immunodeficiency virus (HIV), known uncontrolled hepatitis B infection, active tuberculosis, or severe infection requiring parenteral antibiotic treatment.
* Inadequate hematologic, hepatic and renal function.
* Known second malignancy.
* Impairment of gastrointestinal function.
* Any unstable or clinically significant concurrent medical condition that would, in the opinion of the investigator, jeopardize the safety of a participant, impact their expected survival through the end of the study participation, and/or impact their ability to comply with the protocol.
* History of severe allergic reaction to any of the study intervention components.

The above information was not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (20):
- United States (2):
  - University of California Irvine Medical Center- Site Number : 8400002, Orange, California
  - The University of Texas MD Anderson Cancer Center- Site Number : 8400001, Houston, Texas
- Argentina (4):
  - Investigational Site Number : 0320003, Rosario, Santa Fe Province
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
- Australia (3):
  - Investigational Site Number : 0360002, Sydney, New South Wales
  - Investigational Site Number : 0360001, Woolloongabba, Queensland
  - Investigational Site Number : 0360003, Melbourne, Victoria
- Chile (3):
  - Investigational Site Number : 1520002, Temuco, La Araucanía
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Viña del Mar, Región de Valparaíso
- South Korea (3):
  - Investigational Site Number : 4100002, Seongnam-si, Gyeonggi-do
  - Investigational Site Number : 4100003, Cheongju-si, North Chungcheong
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
- Spain (3):
  - Investigational Site Number : 7240001, Madrid
  - Investigational Site Number : 7240002, Madrid
  - Investigational Site Number : 7240003, Valencia
- Taiwan (2):
  - Investigational Site Number : 1580002, Tainan
  - Investigational Site Number : 1580001, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: TCD16210 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25347&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 20 centers in 7 countries. A total of 95 participants were screened (Part 1: 24; Part 2: 47; Part 3A: 1; Part 4: 23) between 09 June 2020 and 22 December 2022, of which 30 were screen failures.
Pre-assignment Details: The study was conducted in 4 parts (Part 1, 2, 3 and 4), Part 3 was divided into Part 3A and 3B, of which Part 3B was not initiated and no participants were enrolled. The study was terminated due to strategic reasons not related to safety.
Period: Overall Study
Arm/Group | Part 1- SAR442720 140 mg BIW + Pembrolizumab | Part 1- SAR442720 200mg BIW + Pembrolizumab | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%) | Part 3A- SAR442720 100mg BIW + Adagrasib | Part 4- SAR442720 200mg + Pembrolizumab
Started | 4 | 13 | 13 | 19 | 1 | 15
Completed (Here reasons for not completed indicates reasons for treatment discontinuation) | 0 | 0 | 1 | 1 | 0 | 0
Not Completed | 4 | 13 | 12 | 18 | 1 | 15
Not completed — Adverse Event | 0 | 1 | 5 | 3 | 0 | 2
Not completed — Progressive disease | 4 | 11 | 6 | 11 | 1 | 12
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population consisted of participants who took at least 1 dose of any investigational medicinal product (IMP).
Groups:
- Part 1- SAR442720 140mg BIW + Pembrolizumab: Participants were administered SAR442720 140 mg orally BIW on Days 1 and 4 along with pembrolizumab 200 mg via IV infusion Q3W in 21-day cycles until disease progression, unacceptable AEs, or the participant's or investigator's decision to stop the treatment.
- Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%): Participants with PD-L1 TPS>=50% NSCLC were administered SAR442720 200 mg orally BIW on Days 1 and 2 in 21-day cycles along with an IV infusion of pembrolizumab 200 mg on Q3W (21 days cycle) or 400 mg Q6W (42 days cycle) until disease progression, unacceptable AEs, consent withdrawal, or the participant's or investigator's decision to stop the treatment.
- Part 3A- SAR442720 100mg BIW + Adagrasib: Participants were administered SAR442720 100 mg orally BIW on Days 1 and 2 along with adagrasib 400 mg BID in 21-day cycles until disease progression, unacceptable AEs, consent withdrawal, or the participant's or investigator's decision to stop the treatment.
- Total: Total of all reporting groups
Arm/Group | Part 1- SAR442720 140mg BIW + Pembrolizumab | Part 1- SAR442720 200mg BIW + Pembrolizumab | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%) | Part 3A- SAR442720 100mg BIW + Adagrasib | Part 4- SAR442720 200mg + Pembrolizumab | Total
Number analyzed (Participants) | 4 | 13 | 13 | 19 | 1 | 15 | 65
Age, Customized [Count of Participants; unit: Participants]
  From 18 to 64 years | 4 | 6 | 5 | 6 | 1 | 12 | 34
  From 65 to 74 years | 0 | 6 | 3 | 6 | 0 | 3 | 18
  75 years and over | 0 | 1 | 5 | 7 | 0 | 0 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 7 | 7 | 0 | 13 | 39
  Male | 0 | 5 | 6 | 12 | 1 | 2 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 4 | 5 | 5 | 0 | 1 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 2 | 9 | 8 | 14 | 1 | 13 | 47
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: AE: any untoward medical occurrence in participant or clinical study participant, temporally associated with the use of IMP, whether or not considered related to the IMP. TEAEs: AEs that developed or worsened or became serious during treatment-emergent period, defined as time from first administration of IMP (on Day 1) to last administration of IMP + 30 days. SAE: any untoward medical occurrence that, at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was a medically important event.
Time Frame: From first dose of IMP up to 30 days after the last dose; approximately 27 weeks
Population: Safety population consisted of participants who took at least 1 dose of any IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- SAR442720 140mg BIW + Pembrolizumab | Part 1- SAR442720 200mg BIW + Pembrolizumab
Number analyzed (Participants) | 4 | 13
Participants
  TEAEs | 4 | 13
  TESAEs | 0 | 7

2. Primary Outcome: Parts 1 and 3A: Number of Participants With Treatment Related Dose Limiting Toxicities (DLTs)
Description: Potential DLTs were defined as the AEs that occurred during the first cycle (C) of treatment, considered by the investigator to be related to IMP, unless due to disease progression or to a cause obviously unrelated to IMP: Grade(G)>= 4 AEs, G3 neutropenia lasting >7 days or febrile neutropenia; G3 thrombocytopenia with clinically significant bleeding; any G>=3 immune-related AEs; G3 nonhematologic AEs; G3 aspartate transaminase, alanine transaminase, and/or total bilirubin elevations that persist >5 days; possible Hy's law case; G3 QT interval corrected using Fridericia's formula prolongation; retinal vein occlusion any grade; toxicity related to IMP leading to 50% or less dose intensity of SAR442720 and/or delay in initiation of C2 dosing of pembrolizumab by >15 days, in the absence of recovery to baseline or G <=1 AE. Potential DLT were reviewed by Sponsor and investigators to confirm them as DLTs.
Time Frame: Cycle 1 (21 days)
Population: DLT evaluable population consisted of participants who took at least 4 of the 6 planned doses of SAR442720 (Part-1 and Part-3A) and 28 of the 42 planned doses of adagrasib (Part-3A) in the first cycle of the treatment and completed the DLT observation period OR participants who had any DLT observed in the DLT observation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- SAR442720 140mg BIW + Pembrolizumab | Part 1- SAR442720 200mg BIW + Pembrolizumab | Part 3A- SAR442720 100mg BIW + Adagrasib
Number analyzed (Participants) | 4 | 12 | 1
Participants | 0 | 2 | 0

3. Primary Outcome: Part 2: Percentage of Participants With Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a confirmed complete response (CR) or partial response (PR) determined by investigator per response evaluation criteria in solid tumors (RECIST) version 1.1 CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) had reduction in short axis to 10 millimeter (mm) OR disappearance of all nontarget lesions and normalization of tumor marker level. All lymph nodes had nonpathological in size (< 10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. The confidence interval (CI) was estimated using Clopper-Pearson method.
Time Frame: Tumor assessments performed every 9 weeks (56 ±7 days) after the date of first IMP up to end of treatment, approximately 107 weeks
Population: Safety population consisted of participants who took at least 1 dose of any IMP.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%)
Number analyzed (Participants) | 13 | 19
percentage of participants | 23.1 [6.6 to 49.5] | 5.3 [0.3 to 22.6]

4. Primary Outcome: Part 3A: Number of Participants With Treatment-Emergent Adverse Events and Treatment-Emergent Serious Adverse Events
Description: as for outcome 1
Time Frame: From first dose of IMP up to 30 days after the last dose; approximately 7 weeks
Population: Safety population consisted of participants who took at least 1 dose of any IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3A- SAR442720 100mg BIW + Adagrasib
Number analyzed (Participants) | 1
Participants
  TEAEs | 1
  TESAEs | 0

5. Primary Outcome: Part 4: Plasma Concentration of SAR442720 in Combination With Pembrolizumab
Description: Plasma samples were collected at specified timepoints for pharmacokinetic (PK) analysis.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24 hours post-dose on C1 D1, C1 D15, C2 D1; Pre-dose on C1 D8 and C6 D1; end of treatment (Week 45)
Population: PK population consisted of participants who had at least 1 measurable SAR442720 concentration after the first dose. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanogram per milliter (ng/mL)
Arm/Group | Part 4- SAR442720 200mg + Pembrolizumab
Number analyzed (Participants) | 15
nanogram per milliter (ng/mL)
  Pre-dose: C1 D1 | 0 (0)
  0.5 hours post-dose: C1 D1: number analyzed (Participants) | 14
  0.5 hours post-dose: C1 D1 | 207 (376)
  1 hours post-dose: C1 D1: number analyzed (Participants) | 14
  1 hours post-dose: C1 D1 | 262 (323)
  2 hours post-dose: C1 D1 | 342 (324)
  4 hours post-dose: C1 D1 | 488 (200)
  8 hours post-dose: C1 D1: number analyzed (Participants) | 14
  8 hours post-dose: C1 D1 | 492 (220)
  24 hours post-dose: C1 D1: number analyzed (Participants) | 11
  24 hours post-dose: C1 D1 | 272 (94.9)
  Pre-dose: C1 D8: number analyzed (Participants) | 10
  Pre-dose: C1 D8 | 36.5 (23.6)
  Pre-dose: C1 D15: number analyzed (Participants) | 12
  Pre-dose: C1 D15 | 8.67 (21.6)
  0.5 hours post-dose: C1 D15: number analyzed (Participants) | 12
  0.5 hours post-dose: C1 D15 | 458 (524)
  1 hours post-dose: C1 D15: number analyzed (Participants) | 13
  1 hours post-dose: C1 D15 | 629 (615)
  2 hours post-dose: C1 D15: number analyzed (Participants) | 13
  2 hours post-dose: C1 D15 | 757 (441)
  4 hours post-dose: C1 D15: number analyzed (Participants) | 13
  4 hours post-dose: C1 D15 | 649 (267)
  8 hours post-dose: C1 D15: number analyzed (Participants) | 13
  8 hours post-dose: C1 D15 | 540 (226)
  24 hours post-dose: C1 D15: number analyzed (Participants) | 10
  24 hours post-dose: C1 D15 | 342 (127)
  Pre-dose: C2 D1: number analyzed (Participants) | 11
  Pre-dose: C2 D1 | 7.50 (16.7)
  0.5 hours post-dose: C2 D1: number analyzed (Participants) | 11
  0.5 hours post-dose: C2 D1 | 238 (454)
  1 hours post-dose: C2 D1: number analyzed (Participants) | 11
  1 hours post-dose: C2 D1 | 408 (414)
  2 hours post-dose: C2 D1: number analyzed (Participants) | 11
  2 hours post-dose: C2 D1 | 557 (341)
  4 hours post-dose: C2 D1: number analyzed (Participants) | 11
  4 hours post-dose: C2 D1 | 583 (254)
  8 hours post-dose: C2 D1: number analyzed (Participants) | 11
  8 hours post-dose: C2 D1 | 463 (168)
  24 hours post-dose: C2 D1: number analyzed (Participants) | 7
  24 hours post-dose: C2 D1 | 288 (118)
  Pre-dose: C6 D1: number analyzed (Participants) | 3
  Pre-dose: C6 D1 | 21.3 (21.8)
  End of treatment (Week 45): number analyzed (Participants) | 5
  End of treatment (Week 45) | 54.3 (42.5)

6. Primary Outcome: Part 4: Area Under Curve From Zero to Last Concentration Timepoint (AUClast) for SAR442720 Tablets and Capsules
Description: Plasma samples were collected at specified timepoints to determine AUClast for evaluating the impact of food and formulation on the PK of SAR442720 tablet. It was calculated using non-compartmental analysis (NCA) method.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24 hours on C1 D1, C1 D15 and C2D1
Population: PK evaluable population consisted of participants who completed all of C1 and C2D1 with meal information, full PK, and no dose reduction/missed doses on C1D1, C1D15 and C2D1.
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Groups:
- Part 4- SAR442720 200mg Tablet + Pembrolizumab: Participants were administered SAR442720 200 mg orally BIW on Days 1 and 2 in 21-day cycles (as tablet during the first cycle and as capsule from Cycle 2) along with an IV infusion of pembrolizumab 200 mg Q3W (21-day cycle)or 400 mg Q6W (42-day cycle) until disease progression, unacceptable AEs, consent withdrawal, or the participant's or investigator's decision to stop the treatment.
Arm/Group | Part 4- SAR442720 200mg Tablet + Pembrolizumab
Number analyzed (Participants) | 9
hour*ng/mL
  C1 D1 (Tablet/Fed) | 9410 (3310)
  C1 D15 (Tablet/Fasted) | 10800 (4290)
  C2D1 (Capsules/Fasted) | 9800 (3970)

7. Primary Outcome: Part 4: Maximum Observed Plasma Concentration (Cmax) for SAR442720 Tablets and Capsules
Description: Plasma samples were collected at specified timepoints to determine Cmax for evaluating the impact of food and formulation on the PK of SAR442720 tablet. It was calculated using NCA method.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24 hours on C1 D1, C1 D15 and C2 D1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 4- SAR442720 200mg + Pembrolizumab
Number analyzed (Participants) | 9
ng/mL
  C1D1 (Tablet/Fed) | 637 (220)
  C1D15 (Tablet/Fasted) | 828 (310)
  C2D1 (Capsules/Fasted) | 658 (326)

8. Secondary Outcome: Part 1: Plasma Concentration of SAR442720
Description: Plasma samples were collected at specified timepoints for evaluation of SAR442720 PK concentrations.
Time Frame: Pre-dose, 2, 8, hours post-dose on C1 D1 and C2D1; pre-dose C1D8, C1D15, and C6D1; 2 hours C2D2; and end of treatment (Week 22)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1- SAR442720 140mg BIW + Pembrolizumab | Part 1- SAR442720 200mg BIW + Pembrolizumab
Number analyzed (Participants) | 4 | 12
ng/mL
  Pre-dose: C1 D1: number analyzed (Participants) | 3 | 12
  Pre-dose: C1 D1 | 0 (0) | 0 (0)
  2 hours post-dose: C1 D1 | 332 (208) | 519 (270)
  8 hours post-dose: C1 D1: number analyzed (Participants) | 3 | 12
  8 hours post-dose: C1 D1 | 327 (91.0) | 335 (91.0)
  Pre-dose: C1 D8: number analyzed (Participants) | 0 | 8
  Pre-dose: C1 D8 |  | 42.5 (50.4)
  Pre-dose: C1 D15: number analyzed (Participants) | 2 | 8
  Pre-dose: C1 D15 | 267 (328) | 37.1 (25.7)
  Pre-dose: C2 D1: number analyzed (Participants) | 3 | 10
  Pre-dose: C2 D1 | 29.4 (5.40) | 29.6 (24.8)
  2 hours post-dose: C2 D1: number analyzed (Participants) | 3 | 8
  2 hours post-dose: C2 D1 | 516 (145) | 527 (337)
  8 hours post-dose: C2 D1: number analyzed (Participants) | 3 | 8
  8 hours post-dose: C2 D1 | 413 (118) | 409 (205)
  2 hours post-dose: C2 D2: number analyzed (Participants) | 0 | 4
  2 hours post-dose: C2 D2 |  | 698 (350)
  Pre-dose: C6 D1: number analyzed (Participants) | 0 | 1
  Pre-dose: C6 D1 |  | 75.9 (NA) — Standard deviation (SD) cannot be calculated for a single participant.
  End of treatment (Week 22): number analyzed (Participants) | 1 | 4
  End of treatment (Week 22) | 39.0 (NA) — SD cannot be calculated for a single participant. | 221 (334)

9. Secondary Outcome: Part 2: Plasma Concentration of SAR442720
Description: Plasma samples were collected at specified timepoints for evaluation of SAR442720 PK concentrations.
Time Frame: Pre-dose and 2 hours post-dose C1D1 and C2D1; pre-dose on C1D8, C1D15, C6D1; and end of treatment (Week 104)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%)
Number analyzed (Participants) | 12 | 18
ng/mL
  Pre-dose: C1 D1: number analyzed (Participants) | 12 | 16
  Pre-dose: C1 D1 | 0 (0) | 0 (0)
  2 hours post-dose: C1 D1 | 325 (202) | 385 (285)
  Pre-dose: C1 D8: number analyzed (Participants) | 10 | 13
  Pre-dose: C1 D8 | 106 (154) | 100 (172)
  Pre-dose: C1 D15: number analyzed (Participants) | 5 | 8
  Pre-dose: C1 D15 | 149 (234) | 85.1 (81.4)
  Pre-dose: C2 D1: number analyzed (Participants) | 8 | 9
  Pre-dose: C2 D1 | 53.3 (50.8) | 83.9 (159)
  2 hours post-dose: C2 D1: number analyzed (Participants) | 8 | 9
  2 hours post-dose: C2 D1 | 340 (211) | 442 (369)
  Pre-dose: C6 D1: number analyzed (Participants) | 5 | 4
  Pre-dose: C6 D1 | 94.9 (42.8) | 50.1 (16.8)
  End of treatment (Week 104): number analyzed (Participants) | 6 | 5
  End of treatment (Week 104) | 22.3 (39.0) | 19.0 (33.3)

10. Secondary Outcome: Parts 1 and 2: Serum Concentration of Pembrolizumab
Description: Serum samples were collected at specified timepoints for evaluation of pembrolizumab PK concentrations.
Time Frame: Pre-dose and post-dose C1D1; pre-dose on C2D1 and C6D1
Population: PK population consisted of participants who had at least 1 measurable pembrolizumab concentration after the first dose. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1- SAR442720 140mg BIW + Pembrolizumab | Part 1- SAR442720 200mg BIW + Pembrolizumab | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%)
Number analyzed (Participants) | 4 | 10 | 11 | 16
ng/mL
  Pre-dose: C1 D1: number analyzed (Participants) | 2 | 10 | 11 | 16
  Pre-dose: C1 D1 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Post-dose: C1 D1: number analyzed (Participants) | 1 | 7 | 5 | 7
  Post-dose: C1 D1 | 83200 (NA) — SD cannot be calculated for a single participant. | 63600 (11600) | 85200 (38100) | 98900 (55500)
  Pre-dose: C2 D1: number analyzed (Participants) | 4 | 10 | 7 | 8
  Pre-dose: C2 D1 | 15500 (5350) | 14400 (5480) | 10800 (3520) | 9290 (3620)
  Pre-dose: C6 D1: number analyzed (Participants) | 0 | 1 | 6 | 4
  Pre-dose: C6 D1 |  | 46000 (NA) — SD cannot be calculated for a single participant. | 23400 (6450) | 27200 (6350)

11. Secondary Outcome: Parts 1 and 4: Percentage of Participants With Objective Response Rate
Description: ORR was defined as the percentage of participants who had a confirmed CR or PR determined by investigator per RECIST version 1.1 CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) had reduction in short axis to 10 mm OR disappearance of all nontarget lesions and normalization of tumor marker level. All lymph nodes had nonpathological in size (< 10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. The CI was estimated using Clopper-Pearson method.
Time Frame: Tumor assessments performed on C3 D1 (± 7 days) and every 2 cycles up to C7 D1 (± 7 days), and then every 3 cycles thereafter, approximately 23.7 weeks (Part 1), 46 weeks (Part 4)
Population: Safety population consisted of participants who took at least 1 dose of any IMP.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1- SAR442720 140mg BIW + Pembrolizumab | Part 1- SAR442720 200mg BIW + Pembrolizumab | Part 4- SAR442720 200mg + Pembrolizumab
Number analyzed (Participants) | 4 | 13 | 15
percentage of participants | 0 [0.0 to 52.7] | 0 [0.0 to 20.6] | 6.7 [0.3 to 27.9]

12. Secondary Outcome: Part 1: Duration of Response (DoR)
Description: DoR as per RECIST version 1.1 was defined as the interval from the first documentation of CR or PR to the earlier of first documentation of definitive disease progression(PD) or death due to any cause, whichever occurs first. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) had reduction in short axis to 10 mm OR disappearance of all nontarget lesions and normalization of tumor marker level. All lymph nodes had nonpathological in size (< 10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study and the sum must also demonstrate an absolute increase of at least 5 mm. DoR was estimated using Kaplan-Meier method.
Time Frame: Tumor assessments performed on C3 D1 (± 7 days) and every 2 cycles up to C7 D1 (± 7 days), and then every 3 cycles thereafter, approximately 23.7 weeks
Population: Safety population consisted of participants who took at least 1 dose of any IMP and with best overall response (BOR) at least PR. Only responders with BOR with at least a PR were included in the analysis.
Arm/Group | Part 1- SAR442720 140mg BIW + Pembrolizumab | Part 1- SAR442720 200mg BIW + Pembrolizumab
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Part 2: Duration of Response
Description: DoR as per RECIST version 1.1 was defined as the interval from the first documentation of CR or PR to the earlier of first documentation of definitive PD or death due to any cause, whichever occurs first. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) had reduction in short axis to 10 mm OR disappearance of all nontarget lesions and normalization of tumor marker level. All lymph nodes had nonpathological in size (< 10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study and the sum must also demonstrate an absolute increase of at least 5mm. DoR was estimated using Kaplan-Meier method.
Time Frame: as for outcome 3
Population: Safety population consisted of participants who took at least 1 dose of any IMP and with BOR at least PR. Only responders with BOR with at least a PR were included in the analysis.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%)
Number analyzed (Participants) | 3 | 1
months | NA [NA to NA] — NA indicates that the median, upper limit, and lower limit of CI were not estimable due to insufficient number of participants with events. | 16.59 [NA to NA] — NA indicates upper and lower limit of 90% CI was not estimable when only 1 participant was analyzed.

14. Secondary Outcome: Part 2: Number of Participants With Treatment-Emergent Adverse Events and Treatment-Emergent Serious Adverse Events
Description: as for outcome 1
Time Frame: From first dose of IMP up to 30 days after the last dose; approximately 111 weeks
Population: Safety population consisted of participants who took at least 1 dose of any IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%)
Number analyzed (Participants) | 13 | 19
Participants
  TEAEs | 13 | 18
  TESAEs | 9 | 11

15. Secondary Outcome: Part 4: Number of Participants With Treatment-Emergent Adverse Events and Treatment-Emergent Serious Adverse Events
Description: as for outcome 1
Time Frame: From first dose of IMP up to 30 days after the last dose; approximately 50 weeks
Population: Safety population consisted of participants who took at least 1 dose of any IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 4- SAR442720 200mg + Pembrolizumab
Number analyzed (Participants) | 15
Participants
  TEAEs | 15
  TESAEs | 7

16. Secondary Outcome: Part 2: Time to Response (TTR)
Description: TTR was defined as the time interval from the administration of first IMP dose to the first documented evidence of PR or CR determined by the Investigator per RECIST version 1.1. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) had reduction in short axis to 10 mm OR disappearance of all nontarget lesions and normalization of tumor marker level. All lymph nodes had nonpathological in size (< 10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. TTR was estimated using Kaplan-Meier method.
Time Frame: as for outcome 3
Population: as for outcome 13
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%)
Number analyzed (Participants) | 3 | 1
months | 2.23 [2.103 to NA] — NA indicates that the upper limit of CI was not estimable due to insufficient number of participants with events. | 4.34 [NA to NA] — NA indicates upper and lower limit of 90% CI was not estimable when only 1 participant was analyzed.

17. Secondary Outcome: Part 2: Percentage of Participants With Clinical Benefit Rate
Description: Clinical benefit rate was defined as the percentage of participants with confirmed CR or PR at any time or stable disease (SD) of at least 6 months determined by investigator per RECIST version 1.1. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) had reduction in short axis to 10 mm OR disappearance of all nontarget lesions and normalization of tumor marker level. All lymph nodes had nonpathological in size (< 10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. The CI was estimated using Clopper-Pearson method.
Time Frame: as for outcome 3
Population: Safety population consisted of participants who took at least 1 dose of any IMP.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%)
Number analyzed (Participants) | 13 | 19
percentage of participants | 30.8 [11.3 to 57.3] | 21.1 [7.5 to 41.9]

18. Secondary Outcome: Part 2: Percentage of Participants With Disease Control Rate
Description: Disease control rate was defined percentage of participants with confirmed CR or PR or SD as determined by the investigator per RECIST version 1.1. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) had reduction in short axis to 10 mm OR disappearance of all nontarget lesions and normalization of tumor marker level. All lymph nodes had nonpathological in size (< 10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. The CI was estimated using Clopper-Pearson method.
Time Frame: as for outcome 3
Population: Safety population consisted of participants who took at least 1 dose of any IMP.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%)
Number analyzed (Participants) | 13 | 19
percentage of participants | 53.8 [28.7 to 77.6] | 31.6 [14.7 to 53.0]

19. Secondary Outcome: Part 2: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of first IMP administration to the date of the first documented PD determined by the investigator per RECIST version 1.1 or death due to any cause, whichever occurs first. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study and the sum must also demonstrate an absolute increase of at least 5 mm. PFS was estimated using Kaplan-Meier method.
Time Frame: as for outcome 3
Population: Safety population consisted of participants who took at least 1 dose of any IMP.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%)
Number analyzed (Participants) | 13 | 19
months | 3.38 [1.084 to 7.852] | 1.95 [1.117 to 6.111]

20. Secondary Outcome: Part 3A: Plasma Concentration of SAR442720
Description: Plasma samples were collected at specified timepoints for evaluation of SAR442720 PK concentrations. It was calculated using NCA method.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 24 hours post-dose C1D1; pre-dose C1D8; pre-dose, 0.5, 1, 2, 4, 6 post-dose C1D15, and end of treatment (Week 3)
Population: PK population consisted of participants who had at least 1 measurable SAR442720 concentration after the first dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 3A- SAR442720 100mg BIW + Adagrasib
Number analyzed (Participants) | 1
ng/mL
  Pre-dose: C1 D1 | 0 (NA) — SD cannot be calculated for a single participant.
  0.5 hours post-dose: C1 D1 | 0 (NA) — SD cannot be calculated for a single participant.
  1 hours post-dose: C1 D1 | 0 (NA) — SD cannot be calculated for a single participant.
  2 hours post-dose: C1 D1 | 170 (NA) — SD cannot be calculated for a single participant.
  4 hours post-dose: C1 D1 | 432 (NA) — SD cannot be calculated for a single participant.
  6 hours post-dose: C1 D1 | 356 (NA) — SD cannot be calculated for a single participant.
  24 hours post-dose: C1 D1 | 167 (NA) — SD cannot be calculated for a single participant.
  Pre-dose: C1 D8 | 31.5 (NA) — SD cannot be calculated for a single participant.
  Pre-dose: C1 D15 | 36.6 (NA) — SD cannot be calculated for a single participant.
  0.5 hours post-dose: C1 D15 | 34.3 (NA) — SD cannot be calculated for a single participant.
  1 hours post-dose: C1 D15 | 46.6 (NA) — SD cannot be calculated for a single participant.
  2 hours post-dose: C1 D15 | 306 (NA) — SD cannot be calculated for a single participant.
  4 hours post-dose: C1 D15 | 376 (NA) — SD cannot be calculated for a single participant.
  6 hours post-dose: C1 D15 | 310 (NA) — SD cannot be calculated for a single participant.
  End of treatment (Week 3) | 0 (NA) — SD cannot be calculated for a single participant.

21. Secondary Outcome: Part 3A: Plasma Concentration of Adagrasib
Description: Plasma samples were collected at specified timepoints for evaluation of adagrasib PK concentrations. It was calculated using NCA method.
Time Frame: Pre-dose, 1, 2, 4, 6, 8 post-dose C1D1 and C1D15; pre-dose C1D8
Population: PK population consisted of participants who had at least 1 measurable adagrasib concentration after the first dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 3A- SAR442720 100mg BIW + Adagrasib
Number analyzed (Participants) | 1
ng/mL
  Pre-dose: C1 D1 | 0 (NA) — SD cannot be calculated for a single participant.
  1 hours post-dose: C1 D1 | 376 (NA) — SD cannot be calculated for a single participant.
  2 hours post-dose: C1 D1 | 727 (NA) — SD cannot be calculated for a single participant.
  4 hours post-dose: C1 D1 | 1560 (NA) — SD cannot be calculated for a single participant.
  6 hours post-dose: C1 D1 | 1330 (NA) — SD cannot be calculated for a single participant.
  8 hours post-dose: C1 D1 | 1180 (NA) — SD cannot be calculated for a single participant.
  Pre-dose: C1 D8 | 2640 (NA) — SD cannot be calculated for a single participant.
  Pre-dose: C1 D15 | 2110 (NA) — SD cannot be calculated for a single participant.
  1 hours post-dose: C1 D15 | 2150 (NA) — SD cannot be calculated for a single participant.
  2 hours post-dose: C1 D15 | 2910 (NA) — SD cannot be calculated for a single participant.
  4 hours post-dose: C1 D15 | 2880 (NA) — SD cannot be calculated for a single participant.
  6 hours post-dose: C1 D15 | 2510 (NA) — SD cannot be calculated for a single participant.
  8 hours post-dose: C1 D15 | 2320 (NA) — SD cannot be calculated for a single participant.

22. Secondary Outcome: Part 3A: Percentage of Participants With Objective Response Rate
Description: as for outcome 11
Time Frame: Tumor assessments performed till end of treatment, approximately 3 weeks
Population: Safety population consisted of participants who took at least 1 dose of any IMP.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Part 3A- SAR442720 100mg BIW + Adagrasib
Number analyzed (Participants) | 1
percentage of participants | 0 [0.0 to 95.0]

23. Secondary Outcome: Part 3A: Duration of Response
Description: DoR as per RECIST version 1.1 was defined as the interval from the first documentation of CR or PR to the earlier of first documentation of definitive PD or death due to any cause, whichever occurs first. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) had reduction in short axis to 10 mm OR disappearance of all nontarget lesions and normalization of tumor marker level. All lymph nodes had nonpathological in size (< 10 mm short axis). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study and the sum must also demonstrate an absolute increase of at least 5 mm. DoR was estimated using Kaplan-Meier method.
Time Frame: Tumor assessments performed till end of treatment, approximately 3 weeks
Population: as for outcome 13
Arm/Group | Part 3A- SAR442720 100mg BIW + Adagrasib
Number analyzed (Participants) | 0

24. Primary Outcome: Part 4: Time to Reach Maximum Plasma Concentration (Tmax) for SAR442720 Tablets and Capsules
Description: Plasma samples were collected at specified timepoints to determine tmax for evaluating the impact of food and formulation on the PK of SAR442720 tablet. It was calculated using NCA method.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 24 hours on C1 D1, C1 D15 and C2 D1
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | Part 4- SAR442720 200mg + Pembrolizumab
Number analyzed (Participants) | 9
hour
  C1D1 (Tablet/Fed) | 3.75 [1.08 to 24]
  C1D15 (Tablet/Fasted) | 2.02 [0.9 to 7.58]
  C2D1 (Capsules/Fasted) | 3.6 [0.93 to 24]

ADVERSE EVENTS:
Time Frame: Adverse events data was collected from first dose of IMP up to 30 days after the last dose, approximately 27 weeks (Part 1), approximately 111 weeks (Part 2), approximately 7 weeks (Part 3A), and approximately 50 weeks (Part 4). All-cause mortality (death) was collected from first dose of IMP up to end of follow-up, approximately 58 weeks (Part 1), 126 weeks (Part 2), 16 weeks (Part 3A), and 61 weeks (Part 4).
Description: Analysis was performed on safety population.
Arm/Group | Part 1- SAR442720 140mg BIW + Pembrolizumab | Part 1- SAR442720 200mg BIW + Pembrolizumab | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%) | Part 3A- SAR442720 100mg BIW + Adagrasib | Part 4- SAR442720 200mg + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 1/4 | 6/13 | 5/13 | 11/19 | 0/1 | 7/15
Serious Adverse Events (participants affected / at risk) | 0/4 | 7/13 | 9/13 | 11/19 | 0/1 | 7/15
Other Adverse Events (participants affected / at risk) | 4/4 | 13/13 | 12/13 | 16/19 | 1/1 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1- SAR442720 140mg BIW + Pembrolizumab (N=4) | Part 1- SAR442720 200mg BIW + Pembrolizumab (N=13) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%) (N=13) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%) (N=19) | Part 3A- SAR442720 100mg BIW + Adagrasib (N=1) | Part 4- SAR442720 200mg + Pembrolizumab (N=15)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual Impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus Colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 2 (3) | 0 (0) | 0 (0)
Pseudomembranous Colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Tumour Thrombotic Microangiopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central Nervous System Lesion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral Ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Transverse Sinus Thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea At Rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Angiopathy (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1- SAR442720 140mg BIW + Pembrolizumab (N=4) | Part 1- SAR442720 200mg BIW + Pembrolizumab (N=13) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A1 (PDL1 TPS >=50%) (N=13) | Part 2- SAR442720 200mg + Pembrolizumab - Cohort A2 (PDL1 TPS 1% - 49%) (N=19) | Part 3A- SAR442720 100mg BIW + Adagrasib (N=1) | Part 4- SAR442720 200mg + Pembrolizumab (N=15)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 6 (6) | 2 (2) | 5 (7) | 0 (0) | 3 (3)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Ventricular Thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid Irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation Increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 4 (6) | 5 (8) | 0 (0) | 5 (5)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face Oedema (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 3 (4) | 3 (3) | 0 (0) | 3 (3)
Feeling Cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple Organ Dysfunction Syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 3 (3) | 3 (4) | 4 (8) | 0 (0) | 3 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 3 (3) | 3 (4) | 0 (0) | 2 (2)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Temperature Intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 2 (4) | 4 (6) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 3 (3) | 0 (0) | 2 (2) | 3 (5) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Fibrinogen Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Potassium Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Sodium Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection Fraction Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International Normalised Ratio (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International Normalised Ratio Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (10) | 0 (0) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Affective Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic Obstruction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 5 (7) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (4) | 4 (4) | 0 (0) | 2 (2)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angiopathy (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated due to strategic reasons not related to safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT04418661/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT04418661/SAP_001.pdf